CLINICAL TRIAL: NCT06041399
Title: The Effect of Related Blood Markers on Diabetic Peripheral Neuropathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Dbinbin
Record Dates: First submitted 2022-12-26; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Diabetic Peripheral Neuropathy; electromyography; blood parameters

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- diabetic peripheral neuropathy group with hypoglycemic or lipid-lowering drugs. (Experimental): Patients with type 2 diabetic peripheral neuropathy were categorized into the diabetic peripheral neuropathy group with hypoglycemic or lipid-lowering drugs group.The group treated with specific drug,like hypoglycemic or lipid-lowering drugs.
  Interventions: Drug: hypoglycemic Agents(metformin); Drug: lipid-lowering drug(Statin)
- diabetic peripheral neuropathy group without hypoglycemic or lipid-lowering drugs. (No Intervention): Patients with type 2 diabetic peripheral neuropathy were categorized into the diabetic peripheral neuropathy group without hypoglycemic or lipid-lowering drugs group.No hypoglycemic or lipid-lowering drugs were used in this group.
- Diabetic group with hypoglycemic or lipid-lowering drugs. (Experimental): Patients with type 2 diabetes mellitus but not with diabetic peripheral neuropathy were distributed into the Diabetic group with hypoglycemic or lipid-lowering drugs group. group.The group treated with specific drug,like hypoglycemic or lipid-lowering drugs.
  Interventions: Drug: hypoglycemic Agents(metformin); Drug: lipid-lowering drug(Statin)
- Diabetic group without hypoglycemic or lipid-lowering drugs. (No Intervention): Patients with type 2 diabetes mellitus but not with diabetic peripheral neuropathy were distributed into the Diabetic group without hypoglycemic or lipid-lowering drugs group.No hypoglycemic or lipid-lowering drugs were used in this group.

INTERVENTIONS:
Drug: hypoglycemic Agents(metformin) — patients treated with hypoglycemic Agents(metformin)
  Arms: Diabetic group with hypoglycemic or lipid-lowering drugs.; diabetic peripheral neuropathy group with hypoglycemic or lipid-lowering drugs.
Drug: lipid-lowering drug(Statin) — patients treated with lipid-lowering drug(Statin)
  Arms: Diabetic group with hypoglycemic or lipid-lowering drugs.; diabetic peripheral neuropathy group with hypoglycemic or lipid-lowering drugs.

SUMMARY:
The goal of this observational study is to explore the relationship between related blood indicators and diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
This is a multi-center(about five), randomized, double-blind, placebo-controlled clinical trial with over 1000 subjects.Clinical data were collected by consulting the patient's electronic history. The data included demographic information, blood biochemical markers and electromyography. All participants provided their written informed consent to participate in this study.The study protocol was approved by the Ethics Committee of the First Affiliated Hospital of Wenzhou Medical University(KY-2022-R009).

ELIGIBILITY:
Inclusion Criteria:

* patients who had undergone nerve conduction examination by electromyography(EMG).

Exclusion Criteria:

* pregnancy and lactation; chronic liver disease, kidney disease, arrhythmias, malignant diseases, severe respiratory diseases, heart failure, and acute infections;
* patients with alcohol abuse; history of Autoimmune liver disease, liver disease or abnormal liver function at baseline;
* parathyroid diseases (including hyperthyroidism and hypothyroidism);
* pancreatitis, pancreatectomy or any transplant;
* patients with malignancy and any serious concomitant disease limit the existence of life expectancy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2012-02-01 (Actual); Primary Completion 2022-12-18 (Actual); Study Completion 2025-01-02 (Estimated)

PRIMARY OUTCOMES:
the severity of diabetic peripheral neuropathy | From admission to discharge, up to 1 week
  The nerve conduction examination was conducted at a room temperature of 24℃, with the legs warmed using an electric heating pad for at least 10 minutes to achieve a skin temperature of 32-35℃. The nerve conduction velocities and nerve conduction amplitudes were measured for both sides of the upper and lower limbs, including motor and sensory branches of the median nerve; motor and sensory branches of the ulnar nerve; motor branch of peroneal nerve; motor branch of the tibial nerve; sensory branch of the superficial peroneal nerve. In addition, both sides of the tibial nerve F-wave were recorded, and the lower one was regarded as the final F-wave. Slowed/blocked nerve conduction was defined as more than 2.5 standard deviation below the control nerve conduction threshold. Nerve conduction is defined as abnormal when two or more nerve abnormalities are detected.
the presence of diabetic peripheral neuropathy | From admission to discharge, up to 1 week
  When any of the elements of the screening process -- symptoms, signs, or abnormal nerve conduction parameters --was abnormal, medical records would be scrutinized to see if these participants had accepted a previous diabetic peripheral neuropathy diagnosis by a specialist.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China